CLINICAL TRIAL: NCT04347187
Title: Registry Dedicated to Assess the Risk of Ischemic and Hemorrhagic Complications of Long-term Antithrombotic Therapy in Patients With Atrial Fibrillation
Brief Title: REGistry of Long-term AnTithrombotic TherApy-2
Acronym: REGATTA-2
Status: Recruiting | Type: Observational
Sponsor: National Medical Research Center for Cardiology, Ministry of Health of Russian Federation (Other Government)
Responsible Party: Sponsor
Other Study IDs: REGATTA203121975
Record Dates: First submitted 2020-04-10; First posted 2020-04-15 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation, coronary artery disease
MeSH Terms: conditions — Atrial Fibrillation; Coronary Artery Disease | interventions — Anticoagulants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — whole blood, serum, white cells, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Anticoagulants — oral anticoagulants, dual or triple antithrombotic theraphy
  Other Names: antiplatelets

SUMMARY:
To assess the rates of ischemic and hemorrhagic complications of long-term antithrombotic therapy in patients with atrial fibrillation

DETAILED DESCRIPTION:
The register is a Russian prospective single-center observational study of patients who have indications for long-term antithrombotic therapy in connection with atrial fibrillation

ELIGIBILITY:
Inclusion Criteria:

* Documented atrial fibrillation with CHA2DS2VASC > 1

Exclusion Criteria:

* Subjects who are unwilling or unable to provide informed consent. ACS within 12 months before inclusion Severe CHF (NYHA IV) Stroke within 6 months before inclusion Severe liver or muscle disease Severe kidney disease / renal failure with creatinine > 3 mg/dl Conceivable impossibility to come in touch with the patient or his family at 1-year after the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized or outpatients with confirmed atrial fibrillation and CHA2DS2VASC > 1
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2015-01-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
composite of major cardiovascular events | unclusion up to 5 years
  stroke, myocardial infarction, stent thrombosis [definite or probable], or urgent revascularization, cqrdiac death
composite of any bleeding events | unclusion up to 5 years
  major, clinically relevant nonmajor, minor (BARC, ISTH,GARFIELD AF)

SECONDARY OUTCOMES:
Mutations in following genes | inclusion
  CYP2C9*, VKORC1

CONTACTS AND LOCATIONS:
Overall Officials: Elizaveta Panchenko, PhD, Principal Investigator — National Medical Research Center for Cardiology, Ministry of Health of Russian Federation
Locations (1):
- National Medical Research Center for Cardiology, Ministry of Health of Russian Federation, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article after deidentification (text, tables, figures)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 months and ending 36 months following publication
Access Criteria: Researchers who provide a methodologically sound proposal . For individual participant data meta-analysis.

REFERENCES:
- [Background] van Rein N, Heide-Jorgensen U, Lijfering WM, Dekkers OM, Sorensen HT, Cannegieter SC. Major Bleeding Rates in Atrial Fibrillation Patients on Single, Dual, or Triple Antithrombotic Therapy. Circulation. 2019 Feb 5;139(6):775-786. doi: 10.1161/CIRCULATIONAHA.118.036248. PMID 30586754
- [Background] Olsen AS, McGettigan P, Gerds TA, Fosbol EL, Olesen JB, Sindet-Pedersen C, Staerk L, Lock Hansen M, Pallisgaard JL, Kober L, Torp-Pedersen C, Gislason GH, Lamberts M. Risk of gastrointestinal bleeding associated with oral anticoagulation and non-steroidal anti-inflammatory drugs in patients with atrial fibrillation: a nationwide study. Eur Heart J Cardiovasc Pharmacother. 2020 Sep 1;6(5):292-300. doi: 10.1093/ehjcvp/pvz069. PMID 31742339
- [Background] Panchenko E, Kropacheva E, Dobrovolsky A, Titaeva E, Zemlyanskaya O, Trofimov D, Galkina I, Lifshits G, Vereina N, Sinitsin S, Vorobyeva N, Grehova L, Zateyshchikov D, Zotova I, Vavilova T, Sirotkina O, Grontkovskaya A. CYP2C9 and VKORC1 genotyping for the quality of long-standing warfarin treatment in Russian patients. Pharmacogenomics J. 2020 Oct;20(5):687-694. doi: 10.1038/s41397-020-0157-2. Epub 2020 Feb 6. PMID 32024944
- [Background] Kropacheva ES, Khakimova MB, Krivosheeva EN, Zemlyanskaya OA, Panchenko EP. [Severe gastrointestinal bleeding in patients with atrial fibrillation receiving oral anticoagulants (based on REGistry of long-term AnTithrombotic TherApy - REGATTA)]. Ter Arkh. 2021 Sep 15;93(9):1037-1043. doi: 10.26442/00403660.2021.09.201019. Russian. PMID 36286862
- [Background] Mironova Staroverova AI, Panchenko EP, Kropacheva ES, Zemlyanskaya OA. [Resumption of anticoagulant therapy after major bleeding and recurrence of hemorrhagic complications in patients with atrial fibrillation with a high risk of stroke and thromboembolism (based on the results of 20 years of observation)]. Ter Arkh. 2020 Oct 14;92(9):15-23. doi: 10.26442/00403660.2020.09.000655. Russian. PMID 33346426
- [Background] Krivosheeva EN, Panchenko EP, Kropacheva ES, Dobrovolsky AB, Titaeva EV, Mironov VM, Samko AN. Prediction-Determining Outcomes and Their Predictors in Atrial Fibrillation Patients Receiving Multicomponent Antithrombotic Therapy in Real Clinical Practice. Kardiologiia. 2020 Sep 17;60(8):33-45. doi: 10.18087/cardio.2020.8.n1123. PMID 33155957
- [Background] Krivosheeva EN, Kropacheva ES, Panchenko EP, Samko AN. [Thrombotic and hemorrhagic complications in atrial fibrillation patients, undergoing elective percutaneous coronary intervention]. Ter Arkh. 2019 Sep 15;91(9):38-46. doi: 10.26442/00403660.2019.09.000297. Russian. PMID 32598813
- [Background] Kropacheva ES, Zemlyanskaya OA, Krivosheeva EN, Panchenko EP. [Resumption of anticoagulant therapy after major bleeding and the risk of negative events in patients with atrial fibrillation (based on REGistry of Long-term AnTithrombotic TherApy-2 - REGATA)]. Ter Arkh. 2023 Jan 16;94(12):1374-1380. doi: 10.26442/00403660.2022.12.201994. Russian. PMID 37167181
- [Background] Krivosheeva EN, Komarov AL, Panchenko EP, Khakimova MB, Kropacheva ES, Pogorelova OA, Balakhonova TV, Titaeva EV, Dobrovolsky AB, Galyautdinov DM, Vlasova EE. [GDF-15 and the risk of bleeding in patients with stable CAD receiving multicomponent antithrombotic therapy: the results of the prospective REGATA register]. Ter Arkh. 2024 Jul 30;96(7):683-689. doi: 10.26442/00403660.2024.07.202783. Russian. PMID 39106511
- [Background] Kropacheva ES, Zemlyanskaya OA, Panchenko EP. Chronic Kidney Disease is a Predictor of Recurrent Bleeding in Patients With Atrial Fibrillation After Resuming Anticoagulant Therapy (based on REGistry of Long-term AnTithrombotic TherApy (REGATA-2). Kardiologiia. 2023 Nov 8;63(10):55-62. doi: 10.18087/cardio.2023.10.n2284. English, Russian. PMID 37970856